CLINICAL TRIAL: NCT05790746
Title: The Learning Curve for Pure Retroperitoneoscopic Donor Nephrectomy by Using Cumulative Sum Analysis
Brief Title: The Learning Curve for Retroperitoneoscopic Donor Nephrectomy
Status: Completed | Type: Observational
Sponsor: Samsun Liv Hospital (Other)
Responsible Party: Principal Investigator, Mehmet N. Mercimek, MD, FEBU, Associate Professor, MD, FEBU, Samsun Liv Hospital
Other Study IDs: OMU KAEK 11.07.2019/533
Record Dates: First submitted 2023-03-06; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Transplant;Failure,Kidney
Keywords: retroperitoneoscopy; donor nephrectomy; Learning curve; CUSUM analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: The aim of the study is to identify a precise learning curve for pure retroperitoneoscopic donor nephrectomy (RDN).

Methods: Data from 172 consecutive kidney donors who underwent pure RDN between January 2010 and July 2019 were prospectively collected and evaluated. CUSUM (cumulative sum) analysis was used for testing the operation time. Changepoints were determined by using the R program and BinSeg method. The cohort was divided into three groups. Group 1 refers to competence including the first 10 cases, group 2: 11- 48 cases as proficiency, and group 3: the subsequent 124 cases as expert level. Continuous variables were evaluated using one-way ANOVA, and categorical data were evaluated using the Chi-square test

DETAILED DESCRIPTION:
The prospectively collected data of 172 consecutive kidney donors undergoing pure RDN for transplantation at Ondokuz Mayıs University from January 2010 to July 2019 were evaluated retrospectively. Tc-99m mercaptoacetyltriglycine (MAG3) renal scintigraphy was performed to evaluate for split renal function. Three-dimensional computed tomography was performed to evaluate kidney anatomy and vasculature. The final decision for the laterality of surgery was based on the conviction that the better kidney remains with the donor. If both kidneys have equal functional characteristics, the left kidney or the kidney with simpler vascular anatomy was procured based on the transplantation medical review board's decision. The demographic data including age, gender, body mass index (BMI), preoperative renal function, number of renal arteries and veins were recorded. Perioperative variables such as operation time (OT), warm ischemia time (WIT), estimated blood loss (EBL), perioperative and postoperative complications were also recorded. Furthermore, the outcomes of renal recipients including graft function, complications and follow-up were recorded as well. In our previously published article provides a thorough description of the surgical procedure and details for the right and left sides of pure RDN. All RNDs were performed by a single surgeon with experience in retroperitoneoscopic laparoscopic surgery and kidney transplantation.

Learning curve analysis The CUSUM analysis and BinSeg (Binary Segmentation) method Although the CUSUM analysis was first built to evaluate industrial sector performance, it has been adopted in medicine to interpret many surgical techniques learning curve. In a timeline, it calculates the sum of the existing differences between individual operation times and the mean of all operation times. Its main use of in medicine is that calculates the sum of the existing differences between individual operation times and the mean of all operation times in a timeline. The next step is to identify significant change points to determine the development. The "changepoint" package was used in the R program to determine the change points. The changepoints were determined according to the mean variation. BinSeg methods were used to identify two exchange points. Penalty methods were not used to determine surgical time change points. The "Normal" method was used as the test statistic for the surgical time. According to the learning curve analysis methods that are mentioned above, the whole cohort was divided into three groups. Inspired by the Dreyfus model of skill acquisition in the naming of the groups. Thus, group 1 represents competence, group 2 is proficiency level, and group 3 is the expert level.

ELIGIBILITY:
Inclusion Criteria:

* patients with complete data
* patients with consent
* Patients > 18 year-old
* The surgeries performed by the surgeon EO
* Patients who underwent retroperitoneoscopic donor nephrectomy at Ondokuz Mayıs University, Department of Urology

Exclusion Criteria:

* Missing data
* patients without consent
* patients who underwent open of transperitoneal laparoscopic donor nephrectomy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The prospectively collected data of 172 consecutive kidney donors undergoing pure retroperitoneoscopic donor nephrectomy for renal transplantation at Ondokuz Mayıs University, Faculty of Medicine, Department of Urology from January 2010 to July 2019 were evaluated retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-11-03 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Opertaion time | during the surgery (minute)
  From first trocar incision to closure of all incisions
Estimeted blood loss | during the surgery (mL)
  perioperative estimated blood loss
warm ischemia time | during the surgery (second)
  Its starts when the renal artery and vein are controlled and it ends when reperfusion of the graft kidney starts on the back table

SECONDARY OUTCOMES:
Learning curve | through study completion, an average of 1 year
  Number of cases required to achieve reduction in operative time, warm ischemia time, and estimated blood loss.

CONTACTS AND LOCATIONS:
Overall Officials: Ender Ozden, Prof., Study Chair — Ondokuz Mayıs University, Faculty of Medicine
Locations (1):
- Ondokuz Mayıs University, Department of Urology, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pal BC, Modi PR, Rizvi SJ, Chauhan R, Kumar S, Nagarajan R, Kaushal D, Kute VB, Trivedi HL. The Learning Curve of Pure Retroperitoneoscopic Donor Nephrectomy. Int J Organ Transplant Med. 2017;8(4):180-185. Epub 2017 Nov 1. PMID 29321833
- [Result] Kudsi OY, Gokcal F, Bou-Ayash N, Crawford AS. Learning curve of robotic transversus abdominis release in ventral hernia repair: a cumulative sum (CUSUM) analysis. Surg Endosc. 2022 May;36(5):3480-3488. doi: 10.1007/s00464-021-08669-7. Epub 2021 Sep 7. PMID 34494150
- See also: Surgical technique — https://pubmed.ncbi.nlm.nih.gov/32208049/